CLINICAL TRIAL: NCT00508690
Title: Randomized Controlled Trial of Antibiotic Prophylaxis in Elective Laparoscopic Colorectal Surgery: Oral and Systemic Versus Systemic Antibiotics
Brief Title: Trial of Antibiotic Prophylaxis in Elective Laparoscopic Colorectal Surgery: Oral and Systemic Versus Systemic Antibiotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Multinational Trial Organization (Other)
Responsible Party: Principal Investigator, Hiroaki Hata, member, Japan Multinational Trial Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JMTO PREV07-01; UMIN000000776
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Neoplasms
Keywords: Antibiotic Prophylaxis; Colorectal Surgery; Laparoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cefmetazole; Kanamycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV (Active Comparator): Intravenous dose of 1g cefmetazole just before surgery and additional doses every 3hs during surgery
  Interventions: Drug: cefmetazole
- Oral/IV (Active Comparator): 2 doses of oral kanamycin(1g)/ metronidazole(750mg) administration on the day before surgery with intravenous dose of 1g cefmetazole just before surgery and additional doses every 3hs during surgery
  Interventions: Drug: kanamycin/metronidazole

INTERVENTIONS:
Drug: cefmetazole — Intravenous dose of 1g cefmetazole just before surgery and additional doses every 3hs during surgery
  Arms: IV
Drug: kanamycin/metronidazole — 2 doses of oral kanamycin(1g)/ metronidazole(750mg) administration on the day before surgery with intravenous dose of 1g cefmetazole just before surgery and additional doses every 3hs during surgery
  Arms: Oral/IV

SUMMARY:
The purpose of this study is to determine optimal prophylactic antibiotics administration method in elective laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
The use of antibiotic prophylaxis in patients who undergo elective colorectal surgery is now accepted universally. But the rout of administration should be systematic, oral, or both is controversial. Furthermore, although many trails have been performed, no trial limited to laparoscopic surgery is performed. We compare 2 approaches - oral and systemic versus systemic antibiotic prophylaxis - in limited to elective laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal tumor(cancer, adenoma and suspected cases) with planned elective laparoscopic colorectal resection

Exclusion Criteria:

* ECOG Performance Status >=2
* Age<20
* Any organ dysfunction
* Ileus
* Preoperative infectious disease
* Antibiotic administration before surgery
* Steroid administration before surgery
* Neo-adjuvant radiation and/or chemo therapy
* Severe diabetes mellitus
* Pregnancy/lactational woman
* Severe allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence and classification of surgical site infection (SSI) | Within the first 30 days after surgery

SECONDARY OUTCOMES:
Incidence of colitis, other infectious diseases and other postoperative complications. | Within the first 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Hata, MD, Principal Investigator — National Hospital Organization Kyoto Medical Center
Locations (5):
- Japan (5):
  - Kyoto Univercity Hospital, Kyoto, Kyoto
  - National Hospital Organization, Kyoto Medical Center, Kyoto, Kyoto
  - Kyoto Katsura Hospital, Kyoto, Kyoto
  - Tenriyorozu Hospital, Tenri, Nara
  - Kitano Hospital, Osaka, Osaka

REFERENCES:
- See also: UMIN Clinical Trial Registry: Unique trial number UMIN000000776 — http://www.umin.ac.jp/ctr/index.htm